CLINICAL TRIAL: NCT06615570
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single- and Multiple-dose Escalation Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of VX-973 in Healthy Adults
Brief Title: A Phase 1 Dose Escalation Study of VX-973 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX24-973-002
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part A: Single Ascending Dose (Experimental): Participants will be randomized to receive a single dose of VX-973 under fasted conditions.
  Interventions: Drug: VX-973
- Part B: Multiple Ascending Dose (Experimental): Participants will be randomized to receive multiple doses of VX-973 under fasted conditions.
  Interventions: Drug: VX-973
- Placebo Part A (Placebo Comparator): Participants will be randomized to receive placebo matched to VX-973.
  Interventions: Drug: Placebo
- Placebo Part B (Placebo Comparator): Participants will be randomized to receive placebo matched to VX-973.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX-973 — Suspension for oral administration.
  Arms: Part A: Single Ascending Dose; Part B: Multiple Ascending Dose
Drug: Placebo — Suspension for oral administration.
  Arms: Placebo Part A; Placebo Part B

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single and multiple doses of VX-973 in healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (kg/m^2)
* A total body weight of more than (>) 50 kg
* Participants of non-childbearing potential
* Nonsmoker or ex-smoker for at least 3 months before screening

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption, distribution, metabolism, or excretion

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Part A: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day -1 up to Day 30
Part B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day -1 up to Day 85

SECONDARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) of VX-973 | From Day 1 up to Day 30
Part B: Maximum Observed Plasma Concentration (Cmax) of VX-973 | From Day 1 up to Day 85
Part A: Area Under the Concentration Versus Time Curve (AUC) of VX-973 | From Day 1 up to Day 30
Part B: Area Under the Concentration Versus Time Curve (AUC) of VX-973 | From Day 1 up to Day 85
Part A: Time Taken for VX-973 to Reach Maximum Concentration (tmax) | From Day 1 up to Day 30
Part B: Time Taken for VX-973 to Reach Maximum Concentration (tmax) | From Day 1 up to Day 85
Part B: Pain Tolerance Threshold (PTT) for the Cold Pressor Test | From Day 1 up to Day 53

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Salt Lake City, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing